CLINICAL TRIAL: NCT02027376
Title: A Phase Ib Dose Escalation, Open Label, Multicenter Study Evaluating LDE225 (Sonidegib) in Combination With Docetaxel in Triple Negative (TN) Advanced Breast Cancer (ABC) Patients "EDALINE"
Brief Title: Study of LDE225 (Sonidegib) in Combination With Docetaxel in Triple Negative (TN) Advanced Breast Cancer (ABC) Patients
Acronym: EDALINE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2012-12; 2013-001750-96 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2014-01-06 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer; LDE225; Triple Negative; Hormonal Receptor negative; Her2 negative
MeSH Terms: interventions — sonidegib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE225 (sonidegib) plus docetaxel (Experimental): Eligible patients will be included and treated with docetaxel intravenously (75mg/m2)in every three weeks cycles and LDE225 will be administered orally at three dose levels 400, 600 and 800mg QD. Treatment will be repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
  Interventions: Drug: LDE225; Drug: Docetaxel

INTERVENTIONS:
Drug: LDE225
  Other Names: Sonidegib
Drug: Docetaxel
  Other Names: Taxotere

SUMMARY:
This is a single-arm, open-label, phase Ib study. In this trial, patients with Triple Negative (TN) Advanced Breast Cancer (ABC) will be treated with increasing doses of LDE225 (sonidegib) and docetaxel to determine the Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) of the combination.

Eligible patients with hormonal receptors negative and Human Epidermal Growth Factor Receptor 2 (HER2) negative ABC will be included and treated with docetaxel intravenously in every three weeks cycles. LDE225 will be administered orally at three dose levels 400, 600 and 800mg one a day (QD) (a -1 dose level is included just in case dose de-escalation is needed). Treatment will be repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.

The investigators propose to develop a phase Ib trial with the combination of docetaxel with LDE225 in TN ABC patients to define the safety, tolerability and RP2D, as well as to have some information about the efficacy of the combination.

DETAILED DESCRIPTION:
Primary Objective:

To determine the MTD and RP2D of LDE225 administered orally in combination with docetaxel in TN ABC patients.

Primary End-point:

To determine the incidence rate of DLT within the first two cycles of LDE225 in combination with docetaxel at each dose level.

Secondary Objectives:

* To determine the safety and tolerability of LDE225 given in combination with docetaxel.
* To characterize the effects of LDE225 in combination with docetaxel on corrected QT (QTc) intervals and their correlation with systemic drug exposure.
* To evaluate the efficacy of the combination of docetaxel with LDE225 in TN ABC patients.
* To evaluate the Pharmacokinetics (PK) of the combination of docetaxel with LDE225.

Secondary End-points:

* Safety will be assessed by standard clinical and laboratory tests (hematology, serum chemistry). Adverse events grade will be defined by the NCI CTCAE v4.0.
* Changes in QT/QTc from baseline ECG values and correlation with systemic drug exposure.
* The efficacy endpoints are Time To Progression (TTP) and Objective Response Rate (ORR). TTP is measured from the initiation of treatment till disease progression and ORR is defined by RECIST 1.1 criteria as complete response rate + partial response rate.
* The PK will determine whether LDE225 influences the pharmacology of docetaxel. Blood samples will be taken at the times defined in the protocol.

Exploratory Objectives:

* To study potential predictive biomarkers of efficacy by evaluating activation of Hh signaling pathway and related pathways.
* To analyze the pharmacodynamic (PD) treatment effects on the expression of Smo related biomarkers and Hg target genes in correlative samples.
* To correlate biomarker, PD and PK findings with efficacy and toxicity data.

Exploratory End-points:

* Hh gene expression signature associated to pathway activation (at least Shh, Smo, Ptch1, Ptch2, Gli1, Gli2), analyzed in tumor samples.
* Changes in Smo related pathway biomarkers (at least Gli1) in skin and blood correlative samples.
* Pharmacodynamic and biomarker analysis results will be correlated with PK findings, efficacy and toxicity data.

Demographics and Baseline Characteristics:

Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. 95% confidence intervals will be provided for estimates of interest wherever possible.

Safety Analyses:

Adverse events data and serious adverse events will be reported in frequency tables (overall and by intensity). The safety analysis will be performed in the population that has received at least one dose of the drugs.

Efficacy Analyses:

Response will be analyzed in patients with measurable disease that have received at least one dose of the drugs.

TTP will be evaluated in all patients that have received at least one dose of the drugs.

Study population:

Patient with hormonal receptors negative and HER2 negative ABC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is capable to understand and comply with the protocol and has signed the informed consent document.
2. Females with histologically confirmed advanced breast cancer.
3. TN breast cancer by local laboratory determination. Hormonal Receptor (HR) negative defined as < 1% positive cells by Immunohistochemistry (IHC) for both Estrogen Receptor (ER) and Progesterone Receptor (PgR), and HER2 negative defined as in situ hybridization (ISH) negative or IHC 0 or 1+ in the absence of ISH (Note: patients with IHC 2+ must have an ISH determination in order to confirm the HER2 negativity.
4. Measurable or non-measurable disease according to RECIST 1.1 criteria.
5. Patient is at least 18 years of age.
6. World Health Organization (WHO) Performance Status ≤ 1.
7. Life expectancy ≥ 12 weeks.
8. Common laboratory values within normal range (…)
9. A negative serum pregnancy test ≤ 72 hours before starting study treatment for pre-menopausal women and for women < 1 year from the last menstruation date.

Exclusion Criteria:

1. Have received more than 3 prior chemotherapy regimens for ABC.
2. Patients with untreated brain metastases. However, a patient with Central Nervous System (CNS) metastases may participate in this trial if > 4 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable with respect to the tumor at the time of study entry and is not receiving corticosteroid therapy.
3. Patients with acute or chronic liver or renal disease or pancreatitis.
4. Patients with a second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
5. Patients unable to swallow tablets.
6. History of a positive HIV test (HIV testing is not mandatory).
7. History of a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result (Hepatitis B or C testing is not mandatory).
8. Impairment of gastrointestinal (GI) function or GI disease (e.g. ulcerative disease, uncontrolled nausea, vomiting, grade ≥ 2 diarrhea, malabsorption syndrome or small bowel resection).
9. Peripheral vascular disease requiring active therapy or having had surgery < 12 months prior to starting study drug.
10. Impaired cardiac function or clinically significant heart disease (…)

    * A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome
    * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
11. Patients who are receiving treatment with medications that are known to be strong inhibitors or inducers of CYP3A4/5 (listed in Protocol Attachment 3) or drugs metabolized by CYP2B6 or CYP2C9 (listed in Protocol Attachment 3) that cannot be discontinued prior to study entry and for the duration of the study. Medications that are strong CYP3A4/5 inhibitors should be discontinued for at least 2 days, and strong CYP3A4/5 inducers for at least 1 week prior to initiating LDE225 dosing.
12. Patients who have received chemotherapy within a period of time that is < the cycle length used for that treatment (e.g. < 3 weeks for fluorouracil, doxorubicine, epirubicin) prior to starting study drug or who have not recovered from the side effects of such therapy.
13. Patients who have received biologic therapy (e.g. antibodies) ≤ 4 weeks prior to starting study drug or who have not recovered from the side effects of such therapy.
14. Patients who have been treated with a small molecule therapeutic ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy.
15. Patients who have received any other investigational agents ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy.
16. Patients who have received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
17. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin) who cannot discontinue this treatment at least 5 days prior to starting study drug.
18. Patients who are currently receiving immunosuppressive treatment and in whom the treatment cannot be discontinued prior to starting study drug, except in the case of patients with basal cell carcinoma (BCC). Immunosuppressive treatment should be discontinued for at least 1 week prior to initiating LDE225 dosing.

    …

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañón
Locations (5):
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Result] Ruiz-Borrego M, Jimenez B, Antolin S, Garcia-Saenz JA, Corral J, Jerez Y, Trigo J, Urruticoechea A, Colom H, Gonzalo N, Munoz C, Benito S, Caballero R, Bezares S, Carrasco E, Rojo F, Martin M. A phase Ib study of sonidegib (LDE225), an oral small molecule inhibitor of smoothened or Hedgehog pathway, in combination with docetaxel in triple negative advanced breast cancer patients: GEICAM/2012-12 (EDALINE) study. Invest New Drugs. 2019 Feb;37(1):98-108. doi: 10.1007/s10637-018-0614-9. Epub 2018 Jun 9. PMID 29948356
- [Result] Cazet AS, Hui MN, Elsworth BL, Wu SZ, Roden D, Chan CL, Skhinas JN, Collot R, Yang J, Harvey K, Johan MZ, Cooper C, Nair R, Herrmann D, McFarland A, Deng N, Ruiz-Borrego M, Rojo F, Trigo JM, Bezares S, Caballero R, Lim E, Timpson P, O'Toole S, Watkins DN, Cox TR, Samuel MS, Martin M, Swarbrick A. Targeting stromal remodeling and cancer stem cell plasticity overcomes chemoresistance in triple negative breast cancer. Nat Commun. 2018 Jul 24;9(1):2897. doi: 10.1038/s41467-018-05220-6. PMID 30042390
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 patients were enrolled in this trial in the 5 Spanish centers receiving at least one cycle of the combination of oral LDE225 (sonidegib) with intravenous docetaxel. 5 patients were included at Dose Level (DL) 1, 4 patients at DL 2 and 3 patients at DL 3. Two patients at DL 1 and 1 patient at DL 2 were replaced due to early progressive disease.
Pre-assignment Details: Two patients at DL 1 and one patient at DL 2 were replaced due to early progressive disease before completing the first 2 cycles.
Groups:
- LDE225 (Sonidegib) 400mg in Combination With Docetaxel: Cohort 1: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 400mg was administered orally one a day (QD). Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 600mg in Combination With Docetaxel: Cohort 2: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 600mg was administered orally one a day (QD). Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 800mg in Combination With Docetaxel: Cohort 3: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 800mg was administered orally one a day (QD). Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
Period: Overall Study
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Started | 5 | 4 | 3
Completed | 4 | 4 | 3
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LDE225 (Sonidegib) in Combination With Docetaxel: Eligible patients will be included and treated with docetaxel intravenously (75mg/m2) in every three weeks cycles and LDE225 will be administered orally at three dose levels 400, 600 and 800mg QD. Treatment will be repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
  Dose Level 1: 5 patients were included (2 of them were replaced due to progression before completing cycle 2)
  Dose Level 2: 4 patients were included (1 of them were replaced due to progression before completing cycle 2)
  Dose Level 3: 3 patients were included
Arm/Group | LDE225 (Sonidegib) in Combination With Docetaxel
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.25 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 12
Menopausal status [Number; unit: participants]
  Pre-menopausal | 5
  Post-menopausal | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of DLT Within the First Two Cycles of LDE225 (Sonidegib) in Combination With Docetaxel
Description: DLT was defined as the occurrence of any of the following adverse events or abnormal laboratory values (graded according to the NCI-CTCAE version 4.0) assessed as possibly, probably or definitively related to study drugs, occurring within the first two cycles of treatment: Neutropenia grade 4 lasting more than one week, febrile neutropenia, thrombocytopenia grade 3 with bleeding more than grade 2, thrombocytopenia grade 4, Increased plasma creatinine phosphokinase (CK) grade 3-4, any non-hematologic grade 4 toxicity, or grade 3 toxicity except nausea and vomiting, Grade 2 GI toxicity (except nausea and vomiting) lasting more than 2 weeks, Inability to resume dosing for cycles 2 or 3 at the current dose level within 14 days, due to treatment-related toxicity. Dose reductions in cycles 1 and 2 will be considered a DLT
Time Frame: Up to cycle 2
Measure: Count of Participants; unit: Participants
Groups:
- LDE225 (Sonidegib) 400mg in Combination With Docetaxel: Cohort 1: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 400mg was administered orally QD. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 600mg in Combination With Docetaxel: Cohort 2: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 600mg was administered orally QD. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 800mg in Combination With Docetaxel: Cohort 3: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 800mg was administered orally QD. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Number analyzed (Participants) | 5 | 4 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of LDE225 (Sonidegib) in Combination With Docetaxel
Description: MTD was determined by testing increasing doses of LDE225 on dose escalation cohorts 1 to 6 patients. MTD reflects the highest dose tested in which a DLT is experienced by 0 out of 3 or 1 out of 6 patients among the dose levels.
Time Frame: Through study treatment, an average of 2 months
Population: Of the twelve patients included on the study, no Dose Limiting Toxicities (DLTs) were observed at any dose level.
Measure: Number; unit: mg
Groups:
- LDE225 (Sonidegib) in Combination With Docetaxel: Eligible patients were included and treated with docetaxel intravenously (75mg/m2)in every three weeks cycles and LDE225 will be administered orally at three dose levels 400, 600 and 800mg QD. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
Arm/Group | LDE225 (Sonidegib) in Combination With Docetaxel
Number analyzed (Participants) | 12
mg | 800

3. Primary Outcome: Recommended Phase II Dose (RP2D) of LDE225 (Sonidegib) in Combination With Docetaxel
Description: The RP2D was decided by the investigators taken into consideration the information obtained in the study and based on the MTD. To define the RP2D, information about toxicity observed during the full treatment were taken into consideration (relative dose intensity and toxicity observed).
Time Frame: Through study treatment, an average of 2 months
Measure: Number; unit: mg
Groups:
- LDE225 (Sonidegib) in Combination With Docetaxel: Eligible patients will be included and treated with docetaxel intravenously (75mg/m2)in every three weeks cycles and LDE225 will be administered orally at three dose levels 400, 600 and 800mg QD. Treatment will be repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
Arm/Group | LDE225 (Sonidegib) in Combination With Docetaxel
Number analyzed (Participants) | 12
mg | 800

4. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety was assessed by standard clinical and laboratory tests [vital signs including blood pressure, pulse and body temperature, triplicate 12-lead ECGs at screening and on day 1 of cycle 3, blood tests including hematology (hemoglobin, platelets count, red blood cells (RBC), white blood cells (WBC) with differential count and serum chemistry (serum creatinine, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (AP), creatine phosphokinase (CPK))]. Adverse events grade were defined by the NCI CTCAE v4.0.
Time Frame: Through study treatment, an average of 2 months
Measure: Number; unit: number of participants with AE
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Number analyzed (Participants) | 5 | 4 | 3
number of participants with AE | 5 | 4 | 3

5. Secondary Outcome: Changes in QT/QTc From Baseline and Cycle 3 ECG Values.
Description: The QTc intervals have been characterized by comparing QTc at baseline (QTc interval measured in milliseconds (msec) by Fridericia's formula) and at cycle 3 pre-dose, 1 hour post-dose, 2 hours post-dose, 4 hours post-dose and 6 hours post-dose.
Time Frame: From baseline to cycle 3
Population: Only 6 patients received cycle 3. Results are shown from the predose, at 1 hour and 2 hours post-dose for 6 patients and at 4 hours and 6 hours post-dose for 5 patients.
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | LDE225 (Sonidegib) in Combination With Docetaxel
Number analyzed (Participants) | 6
milliseconds
  Cycle 3, Predose | 28.5 [-26 to 82.5]
  Cycle 3, 1 hour | 4.5 [-15 to 23.8]
  Cycle 3, 2 hours | 9.5 [-5.2 to 24.3]
  Cycle 3, 4 hours: number analyzed (Participants) | 5
  Cycle 3, 4 hours | 2.8 [-23 to 29.1]
  Cycle 3, 6 hours: number analyzed (Participants) | 5
  Cycle 3, 6 hours | 4.3 [-15 to 23.2]

6. Secondary Outcome: Time To Progression (TTP)
Description: Tumor assessments were performed until disease progression in order to evaluate the TTP. TTP is defined as the time from the date of the first dose to the first date of objectively determined progressive disease. For patients not known to have objectively-determined progressive disease, TTP will be censored at the date of the last objective progression-free assessment. For patients who receive subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression, TTP will be censored at the date of last objective progression-free assessment prior to the initiation of postdiscontinuation systemic anticancer therapy.
Time Frame: Through study treatment, an average of 2 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Number analyzed (Participants) | 5 | 4 | 3
days | 42.0 [29 to 84] | 42.5 [20 to 64] | 188 [155 to NA] — The upper limit of the Confidence Interval (CI) from LDE225 800mg was censored due to one patient discontinued the study treatment due to toxicity and was on Complete Response (CR).

7. Secondary Outcome: LDE225 (Sonidegib) Trough Concentration (Pharmacokinetics (PK))
Description: To evaluate the effect of LDE225 on the docetaxel PK, the main pharmacokinetic parameters of docetaxel were estimated on Day 1 of Cycles 1 and 2 of treatment, and compared between them. PK parameters were estimated by non-compartmental approach using Phoenix® WinNonlin® software (version 7.0). In the case of the effect of docetaxel on the LDE225 PK, since patients were always under both drugs at all the assessed PK profiles, the trough LDE225 concentrations obtained in our study were compared with those simulated from a previous developed PK model from LDE225 given as monotherapy. Therefore, a population PK model of LDE225 reported in the literature and developed in healthy subjects and patients with advanced solid tumors was implemented in NONMEN version 7.3 program and Monte-Carlo simulations of LDE225 concentrations after the same doses than those of our study, were performed.
Time Frame: Up to cycle 2
Population: At LDE225 600 mg, one patient was discontinued after first cycle.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Number analyzed (Participants) | 5 | 3 | 3
mg/L | 0.398 (0.335) | 0.392 (0.086) | 0.727 (0.539)

8. Secondary Outcome: Docetaxel Clearance on Cycle 1 and Cycle 2 (Pharmacokinetics (PK))
Description: PK sampling of docetaxel was performed on Day 1 of Cycle 1 and 2 of treatment and docetaxel concentrations. Blood samples were collected into ethylenediaminetetraacetic acid (EDTA) K3 tubes and after plasma separation by centrifugation were stored at -70 degrees Celsius until analysis.
Time Frame: Cycles 1 and 2
Population: At LDE225 600 mg, one patient was discontinued after first cycle.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | LDE225 (Sonidegib) in Combination With Docetaxel
Number analyzed (Participants) | 11
L/h
  Cycle 1 Day 1 | 48.8 (19.6)
  Cycle 2 Day 1 | 42.7 (27.8)

9. Secondary Outcome: Objective Response Rate (ORR)
Description: Tumor response was assessed using RECIST 1.1 criteria. The best response across all treatment was recorded. ORR is defined as the percentage of patients with a complete or partial response out of the patients who had measurable disease at baseline.
Time Frame: Through study treatment, an average of 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
Number analyzed (Participants) | 5 | 3 | 2
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Through study treatment, average of 2 months
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation of study treatment.
Groups:
- LDE225 (Sonidegib) 400mg in Combination With Docetaxel: Cohort 1: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 400mg was administered orally one a day. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 600mg in Combination With Docetaxel: Cohort 2: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 600mg was administered orally one a day. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
- LDE225 (Sonidegib) 800mg in Combination With Docetaxel: Cohort 3: Eligible patients were included and treated with docetaxel intravenously (75mg/m2) in every 3 weeks cycles and LDE225 800mg was administered orally one a day. Treatment was repeated on day 1 of a 21-day cycle until radiographic or symptomatic progression, unacceptable toxicity or withdraws informed consent.
Arm/Group | LDE225 (Sonidegib) 400mg in Combination With Docetaxel | LDE225 (Sonidegib) 600mg in Combination With Docetaxel | LDE225 (Sonidegib) 800mg in Combination With Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDE225 (Sonidegib) 400mg in Combination With Docetaxel (N=5) | LDE225 (Sonidegib) 600mg in Combination With Docetaxel (N=4) | LDE225 (Sonidegib) 800mg in Combination With Docetaxel (N=3)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Overdose of grade 1. This patient took 800mg once instead of 600mg (only took one additional tablet) during cycle 3 at DL 2. No any additional AEs were observed due to this intake of a higher dose of sonidegib.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 (Sonidegib) 400mg in Combination With Docetaxel (N=5) | LDE225 (Sonidegib) 600mg in Combination With Docetaxel (N=4) | LDE225 (Sonidegib) 800mg in Combination With Docetaxel (N=3)
Fatigue (General disorders) | 2 | 2 | 2 — Grade 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 — Grade 1
Anemia (Blood and lymphatic system disorders) | 4 | 1 | 1 — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 — Grade 2
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 — Grade 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 2 — Grade 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 — Grade 1
Alkaline Phosphatase increased (Investigations) | 2 | 1 | 1 — Grade 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 — Grade 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 — Grade 1
Neutrophil count decreased (Investigations) | 1 | 0 | 2 — Grade 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 1 — Grade 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 — Grade 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 — Grade 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 — Grade 4
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 — Grade 2
White blood cell decreased (Investigations) | 0 | 2 | 0 — Grade 1
White blood cell decreased (Investigations) | 0 | 1 | 0 — Grade 2
White blood cell decreased (Investigations) | 0 | 0 | 1 — Grade 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 — Grade 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 — Grade 3
Creatine Phosphokinase (CPK) increased (Investigations) | 0 | 0 | 1 — Grade 3
Fatigue (General disorders) | 1 | 0 | 1 — Grade 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 — Grade 2
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 1 — Grade 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 — Grade 2
Phlebitis (Vascular disorders) | 0 | 0 | 1 — Grade 2
Neutrophil count decreased (Investigations) | 1 | 1 | 0 — Grade 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 — Grade 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0 — Grade 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Grade 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 — Grade 1
Creatine Phosphokinase (CPK) increased (Investigations) | 0 | 1 | 0 — Grade 1
Creatinine increased (Investigations) | 0 | 1 | 0 — Grade 1
Paronychia (Infections and infestations) | 0 | 1 | 0 — Grade 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 — Grade 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 — Grade 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 — Grade 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 — Grade 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Grade 1
Eyelid function disorder (Eye disorders) | 0 | 0 | 1 — Grade 1
Photophobia (Eye disorders) | 0 | 0 | 1 — Grade 1
Watering eyes (Eye disorders) | 0 | 0 | 1 — Grade 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Grade 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less